CLINICAL TRIAL: NCT03009760
Title: A Phase I , Study to Investigate Pharmacokinetics and Pharmacodynamics of Single and Multiple Dose of CJ-12420 50mg, 100mg in Helicobacter Pylori ?
Brief Title: To Investigate Pharmacokinetics and Pharmacodynamics of CJ-12420 After Single and Multiple Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [CJ_APA_104]
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CJ-12420 50mg(HP-) (Experimental): CJ-12420 50mg in H. pylori negative subject
  Interventions: Drug: CJ-12420 50mg(HP-)
- CJ-12420 100mg(HP-) (Experimental): CJ-12420 100mg in H. pylori negative subject
  Interventions: Drug: CJ-12420 100mg(HP-)
- CJ-12420 50mg(HP+) (Experimental): CJ-12420 50mg in H. pylori positive subject
  Interventions: Drug: CJ-12420 50mg(HP+)
- CJ-12420 100mg(HP+) (Experimental): CJ-12420 100mg in H. pylori positive subject
  Interventions: Drug: CJ-12420 100mg(HP+)

INTERVENTIONS:
Drug: CJ-12420 50mg(HP-) — CJ-12420 50mg in H. pylori negative subject
  Other Names: not yet determined
  Arms: CJ-12420 50mg(HP-)
Drug: CJ-12420 100mg(HP-) — CJ-12420 100mg in H. pylori negative subject
  Other Names: not yet determined
  Arms: CJ-12420 100mg(HP-)
Drug: CJ-12420 50mg(HP+) — CJ-12420 50mg in H. pylori positive subject
  Other Names: not yet determined
  Arms: CJ-12420 50mg(HP+)
Drug: CJ-12420 100mg(HP+) — CJ-12420 100mg in H. pylori positive subject
  Other Names: not yet determined
  Arms: CJ-12420 100mg(HP+)

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and pharmacodynamics of CJ-12420 after single and multiple dose administration according to H. pylori infection.

DETAILED DESCRIPTION:
1. Cohort 1: To investigate the pharmacokinetics and pharmacodynamics of CJ-12420 after the multiple dose administration in H. pylori negative volunteers.
2. Cohort 2: To investigate the pharmacokinetics and pharmacodynamics of CJ-12420 after the single dose administration in H. pylori positive volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 20 to 45 years of age (inclusive)
* Body mass index (BMI) in the range of 19~28 kg/㎡ and weighted at least 50kg
* Medically healthy with no clinically significant vital signs (blood pressure in the sitting position, pulse rate)

  * 90 mmHg ≤ systolic blood pressure ≤ 140 mmHg
  * 50 mmHg ≤ diastolic blood pressure ≤ 95 mmHg
  * 45 beats per minute ≤ pulse rate ≤ 95 beats per minute
* Understood the requirements of the study and voluntarily consented to participate in the study
* Agreed to be sexually abstinent or to use a condom or spermicide when engaging in sexual activity and not to donate sperm during the course of the study for 30 days following completion of the study
* Non-smokers or non-users of nicotine-containing products for at least 1 year
* [Cohort 1] H. pylori negative as determined by urea breath test and serum IgG antibody
* [Cohort 2] H. pylori positive as determined by urea breath test and serum IgG

Exclusion Criteria:

* History of clinically significant gastrointestinal, renal, hepatic, neurologic, hemato-oncologic, endocrine, pulmonary, immunologic, psychiatric, musculoskeletal, or cardiovascular disease or any other condition, which in the opinion of the investigators, would jeopardize the safety of the subject or impact the validity of the study results
* History of allergy or hypersensitivity to any drug, including prior serious adverse reaction to PPIs or P-CABs
* Undergone surgery or in a medical condition, which in the judgment of the PI or investigators may affect absorption, distribution, metabolism or elimination of the study drug
* Administered other drug(s) in other clinical study within 60 days prior to screening visit
* Donated blood within 60 days or blood components within 30 days, or had been transfused plasma within 30 days prior to screening visit
* On special diet or have experienced substantial changes in eating habits within 30 days prior to screening visit
* Used any prescription medication within 14 days, or any other OTC medications including herbal products within 7 days prior to screening visit
* Consumed over 21 units/week of alcohol
* Consumed over 5 units/day of caffeine-containing beverage
* Positive urine screen for drugs and/or cotinine
* Positive blood screen for human immunodeficiency virus (HIV), hepatitis B or C, or syphilis
* Clinically significant abnormalities of liver function tests (≥1.5 fold of normal upper limit in the level of L-alanine aminotransferase (ALT), L-aspartate aminotransferase (AST) or total bilirubin)
* Unable to bear pH meter catheter insertion
* History of symptomatic GERD, erosive esophagitis, duodenal ulcer, gastric ulcer, Barrett's esophagus, or Zollinger-Ellison syndrome
* Clinically significant observations considered as unsuitable based on medical judgment by investigators

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of CJ-12420 | up to 12 hours

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of CJ-12420 | up to 12 hours
Time of maximum observed concentration(tmax) of CJ-12420 | up to 12 hours
Half life(t1/2β) of CJ-12420 | up to 12 hours
Mean pH | Day -1, Day 1, Day 7 up to 24 hours
  Data from the pH probe monitoring
Time at pH > 4(%) | Day -1, Day 1, Day 7 up to 24 hours
  the percent of time the pH as data from the pH probe monitoring
Time at pH > 6(%) | Day -1, Day 1, Day 7 up to 24 hours
  the percent of time the pH as data from the pH probe monitoring

IPD SHARING:
Plan to Share IPD: No